CLINICAL TRIAL: NCT00275522
Title: A Randomized Open-label Study to Compare the Safety and Efficacy of Two Different Sirolimus Regimens With a Tacrolimus + Mycophenolate Mofetil Regimen in De Novo Renal Allograft Recipients.
Brief Title: The Comparison of Three Different Immunosuppressant Regimens in Kidney Transplant Recipients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Mark D. Stegall, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1302-04
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus

SUMMARY:
The study is being done to compare the safety and effects (good and bad) of three different combinations of immunosuppression drugs used by kidney transplant recipients while also looking at their kidney function.

DETAILED DESCRIPTION:
This is an open-label, randomized, comparative, multinational study. The study will be looking at the kidney function of kidney transplant recipients, while also comparing the safety and the effects (good and bad) of three different combinations of immunosuppression drugs in combination with prednisone, following treatment with Daclizumab (Zenapax). The three combinations are; (1) sirolimus and tacrolimus followed by the withdrawal of tacrolimus after three months; (2) sirolimus and mycophenolate mofetil (MMF); and (3) tacrolimus and MMF. The participants will be required to return to throughout the next 24 months following their transplant for physical exams, chest x-ray, blood, and urine tests. Participants will be put into one of three groups, and receive the study drugs starting on the day of transplant. Due to some drugs affecting the drug levels of sirolimus, participants need to agree not to take any new drugs during the study unless approved by the study doctor.

ELIGIBILITY:
Participants must be at least between the ages of 18 and 75, and will be receiving their first or second kidney transplant.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Calculated creatinine clearance at 12 months after transplantation.

SECONDARY OUTCOMES:
Calculated creatinine clearance at 26, 78, and 104 weeks post transplantation.
Serum creatinine at 26, 52, 78, and 104 weeks post transplantation.
Subject and graft survival at 26, 52, 78, and 104 weeks post transplantation.
Incidence and severity of biopsy-confirmed acute rejection at 26, 52, 78, and 108 weeks post transplantation.
Severity of rejection, including histological grade of the first acute rejection episode.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Stegall, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States